CLINICAL TRIAL: NCT04572256
Title: MOntelukast as a Potential CHondroprotective Treatment Following Anterior Cruciate Ligament Reconstruction (MOCHA Trial)
Acronym: MOCHA
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Austin V Stone (Other)
Collaborators: Duke University (Other); The Cleveland Clinic (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Austin V Stone, Director of Research Orthopedic Surgery, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 60266
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: ACL Injury; Meniscus Tear; Post-traumatic Osteoarthritis
Keywords: knee ligament; osteoarthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Montelukast (Experimental): Patients will receive oral montelukast (10 mg) daily for 6 months after surgery.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Patients will receive an oral placebo daily for 6 months after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — The novel use of oral montelukast offers the potential of a disease modifying treatment to prevent irreversible cartilage loss after ACL injury. 10mg of oral Montelukast will be taken daily for 6 months post surgery.
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — An oral placebo will be taken daily for 6 months post surgery.
  Arms: Placebo

SUMMARY:
This is a multicenter randomized, placebo-controlled trial to assess whether a 6-month course of oral montelukast after ACL reconstruction reduces systemic markers of inflammation and biochemical and imaging biomarkers of cartilage degradation. This study will specifically target older ACL reconstruction patients with concomitant meniscal injuries as this group is at greatest risk of rapid PTOA progression. Patients will randomly be assigned to receive oral montelukast (10 mg) versus placebo daily for 6 months after surgery.

DETAILED DESCRIPTION:
After anterior cruciate ligament (ACL) reconstruction, patient-reported outcomes are improved 10 years post-surgery. Cytokine concentrations, however, remain elevated years after surgery; over 80% of patients with combined ACL and meniscus injuries have post-traumatic osteoarthritis (PTOA) within 10-15 years after injury. Since pain nociceptors are not located in the articular cartilage, patient-reported outcomes improve despite progressive, irreversible cartilage loss, thus making PTOA a "silent killer." Because early cartilage loss progresses without pain and dysfunction, the prevalence of PTOA continues to increase. PTOA now represents the most common cause of military disability.

Our recent results illustrate the downstream cytokine and degradative enzyme activity following ACL reconstruction. ACL and meniscus injury initiate a biochemical cascade resulting in cartilage degradation and this process involves an up-regulated pro-inflammatory response with a dysregulated anti-inflammatory response. Single-dose intra-articular anti-inflammatory treatment appears to reduce hyaline cartilage degradation shortly after the time of injury based on synovial fluid measures of type II collagen degradation. The intra-articular inflammatory milieu at the time of surgery appears to predict the patient symptom state two years later; however, the effectiveness of preoperative anti-inflammatory treatments in impacting patient symptoms or slowing long-term PTOA progression is as yet unclear. A lack of efficacy in preoperative interventions may be attributed to a profound inflammatory stimulus from surgical reconstruction of the ACL. The postoperative inflammatory cascade results in articular cartilage and meniscus degradation due to matrix degrading enzymes, especially those which breakdown type II collagen.

PTOA affects the whole joint organ including the cartilage, synovium, and bone. PTOA progression is multifaceted and includes activation of the pro-inflammatory Nuclear Factor Kappa-B (NFkB) pathway, an increase in pro-inflammatory M1 macrophages, cell senescence, and bone remodeling. Limiting the biochemical cascade through an innovative disease modifying treatment to target upstream activity will potentially treat all components of the knee, thereby lessening the inflammatory response, reducing cartilage catabolism, and potentially improving pathologic bony remodeling observed after ACL reconstruction. The early proteomic PTOA response is more similar to inflammatory rheumatoid arthritis than idiopathic OA; thus, long-acting agents which better regulate pro-inflammatory cytokine activity may more successfully limit tissue destruction. By re-purposing approved therapeutics with proven immune efficacy, a readily-available and cost-effective strategy for disease modification may be possible.

Montelukast was first approved for clinical use in 1998 for prophylaxis and chronic treatment of asthma. The drug selectively inhibits the cysteinyl leukotriene receptor 1 (CysLT1). Montelukast blocks the actions of cysteinyl leukotriene D4 (LTD4), which is produced through the arachidonic acid pathway. This pro-inflammatory signal is released from several cells including the inflammatory mast cells and eosinophils. Montelukast also appears to address multiple PTOA mechanisms by inhibiting cysteinyl leukotrienes. Cysteinyl leukotriene inhibition in animal and laboratory models of PTOA resulted in the elimination of senescent cells, reduced NFkB activation, decreased concentrations of pro-inflammatory and catabolic factors and reactive oxygen species (ROS) while increasing expression of anti-inflammatory factors (inducing anti-inflammatory M2 macrophage infiltration), inhibiting osteoclastogenesis and improving bone quality. The novel use of oral montelukast offers the potential of a disease modifying treatment to prevent irreversible cartilage loss after ACL injury.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing primary ACL reconstruction
2. Age between 25-50
3. Concomitant meniscus injury

Exclusion Criteria:

1. Undergoing revision procedures
2. Multiple ligament injuries requiring multiple ligament reconstruction/repair
3. Depressive symptoms and/or those who endorse suicidal ideation at the time of enrollment (PHQ-9 score >= 15)
4. Found to not have a meniscus tear at the time of surgery

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Serum prostaglandin E2 | Change between Visit 3 (10 days post surgery) and Visit 6 (1 year post surgery)
  Prostaglandin E2 is a potential inflammatory mediator, and it is being measured to directly assess whether treatment reduces this systemic inflammatory marker. Greater serum prostaglandin is associated with greater inflammation.
T1rho relaxation time on MRI | Change between Visit 4 (4 weeks post surgery) and Visit 6 (1 year post surgery)
  T1rho relaxation time is a validated measure of proteoglycan content within the cartilage, and can be assessed on MRI. Increased T1rho relaxation time is associated with increased cartilage degeneration.
Shape of the medial femoral condyle on MRI | Change between Visit 4 (4 weeks post surgery) and Visit 6 (1 year post surgery)
  The shape of the medial femoral condyle has been previously demonstrated to change after ACL reconstruction and is predictive of later cartilage changes. Flattening and widening of the medial femoral condyle are considered to be indicative of later cartilage changes.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Change between Visit 3 (10 days post surgery) and Visit 6 (1 year post surgery)
  The KOOS is a patient-reported outcome instrument that is comprised of 5 subscales (Pain, Symptoms, Activities of Daily Living, Sports and Recreation, and Quality of Life) with each scale being scored from 0 to 100 with higher scores being indicative of a superior outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Stone, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- UK Healthcare at Turfland, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobs CA, Conley CEW, Kraus VB, Lansdown DA, Lau BC, Li X, Majumdar S, Spindler KP, Lemaster NG, Stone AV. MOntelukast as a potential CHondroprotective treatment following Anterior cruciate ligament reconstruction (MOCHA Trial): study protocol for a double-blind, randomized, placebo-controlled clinical trial. Trials. 2022 Jan 31;23(1):98. doi: 10.1186/s13063-021-05982-3. PMID 35101085